CLINICAL TRIAL: NCT01057134
Title: Cutera UHAIR for Hair Removal
Brief Title: Ultrasound Device for Hair Removal
Status: Completed | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-09-UP01; C-09-UP01 (Other: Cutera Inc.)
Record Dates: First submitted 2010-01-25; First posted 2010-01-27 (Estimated); Results first posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Hair Removal
Keywords: Hair Reduction Arm Leg; Unwanted hair

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Site treated with UHAIR (Experimental): The arm, calf, and thigh will be treated
  Interventions: Device: Cutera Ultrasound Device

INTERVENTIONS:
Device: Cutera Ultrasound Device — Pulse duration 10-100 ms, fluence greater or equal to 50 J/cm2, contact tip temperature 5-30 celsus, frequency 5-20 MHz.
  Other Names: UHAIR

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the Cutera UHAIR ultrasound device for hair removal.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the Cutera UHAIR device for safety and efficacy for removal and long term reduction of unwanted hair on subjects with Fitzpatrick skin types I-IV and dark (black or brown), red, and blonde colored hair.

At investigator's discretion, each subject will receive treatments and will be scheduled for follow-up visits after the final treatment. The treated area(s) will be photographed at each visit for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age
* Fitxpatrick skin type I-IV
* Area with unwanted hair
* Subject must be able to read, understand and sign the consent form
* Subject must adhere to the follow-up schedule and study instruction

Exclusion Criteria:

* Simultaneous participation in any other clinical study
* Inability or unwillingness to follow the treatment schedule
* Inability or unwillingness to sign the informed consent
* Infection in the target area
* Any disease or condition that could impair wound healing
* History of keloid formation
* History of malignant tumors in the target area
* Skin abnormalities in the target area, e.g. cuts, scrapes, wounds, scars, large moles
* History of hair removal in target area (light based or electrolysis)
* Pregnant or lactating

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Subjects were treated on the calf, thigh, and arm with the Cutera UHAIR device.
Period: Overall Study
Arm/Group | All Study Participants
Started | 10
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Hair Count in the Treated Area
Description: Percent hair reduction 3 months post final treatment compared to baseline in the treated areas
Time Frame: baseline and 3 months post final treatment (up to 28 weeks)
Measure: Mean (Standard Deviation); unit: percentage of hair reduction
Arm/Group | Arms | Calf | Thigh
Number analyzed (Participants) | 9 | 9 | 9
percentage of hair reduction | 13.1 (9.1) | 10.7 (9.9) | 18.7 (15.5)

ADVERSE EVENTS:
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Study Participants (N=10)
Blistering (Skin and subcutaneous tissue disorders) | 2
Discomfort (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No